CLINICAL TRIAL: NCT07103421
Title: Effect of Non-Surgical Periodontal Therapy on Cystatin C Levels in Healthy and Renal Impaired Patients
Brief Title: Impact of Non Surgical Periodontal Therapy on Cystatin C Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Tishreen U _ periodontic
Record Dates: First submitted 2025-07-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis, Chronic Kidney Disease
Keywords: Non-Surgical Periodontal Therapy, Cystatin C, periodontis, Renal biomarkers
MeSH Terms: conditions — Periodontitis; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Three parallel groups: healthy controls, periodontis patients without systemic disease, and periodontis patients with chronic kidney disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy controls (No Intervention): 10 systemically and periodontally healthy patients who will not receive any periodontal treatment. Cystatin C levels will be measured at baseline.
- Periodontitis patients (Experimental): 10 patients with periodontitis but no systemic diseases who will receive Non-Surgical Periodontal Therapy (scaling and root plannong). Cystatin C levels will be measured before and after treatment.
  Interventions: Diagnostic Test: Non-Surgical Periodontal Therapy
- Periodontitis with CKD (Experimental): 10 patients with periodontitis and 1-3 chronic kidney disease who will receive non-surgical periodontal therapy. Cystatin C levels and renal function will be monitored.
  Interventions: Diagnostic Test: Non-Surgical Periodontal Therapy

INTERVENTIONS:
Diagnostic Test: Non-Surgical Periodontal Therapy — Non-surgical periodontal therapy involves the removal of bacterial plaque and calculus from tooth surfaces and root surfaces beneath the gum line using manual or ultrasonic instruments. This treatment is performed for patients with periodontitis to improve gum health and reduce inflammation. Serum cystatin C levels will be compared before and after treatment between healthy patients and those with renal impairment.
  Arms: Periodontitis patients; Periodontitis with CKD

SUMMARY:
Study the effect of non-surgical periodontal therapy on cystatin C levels in gingival crevicular fluid and serum in both healthy patients and patients with renal impairment. The number of participants is 30 individuals, divided into three groups receiving conservative periodontal treatment (scaling and root planing):Systemically and periodontally healthy patients, Patients with periodontitis without systemic diseases, and Patients with periodontitis and chronic kidney disease. The study also aims to determine the relationship between the severity of periodontal disease and kidney function by measuring cystatin C levels, which is an important biomarker for both conditions. Additionally, it seeks to assess whether non-surgical periodontal therapy can be included in the treatment protocols for kidney patients to improve their quality of life.

DETAILED DESCRIPTION:
Periodontal diseases, particularly gingivitis and periodontitis, are common inflammatory conditions affecting the tooth-supporting tissues. These diseases induce both local and systemic inflammatory responses, which may impact other organs, including the kidneys. Cystatin C (CSTC) is an inhibitor of cysteine proteases and is considered an important biomarker for kidney function, as its serum levels rise in cases of renal impairment. Periodontal diseases may contribute to elevated serum cystatin C levels due to systemic inflammation caused by bacterial infection and inflammatory mediators circulating in the bloodstream. On the other hand, non-surgical periodontal therapy (e.g., scaling and root planing) may reduce both local and systemic inflammation, potentially improving cystatin C levels and kidney function. This study aims to: Assess and compare cystatin C levels in serum and gingival crevicular fluid (GCF) among healthy individuals and patients with periodontitis، Examine the effect of non-surgical periodontal therapy on serum and GCF cystatin C levels in patients with renal impairment compared to healthy controls، and Analyze the relationship between periodontitis severity and kidney function by correlating cystatin C levels with other renal markers (e.g., glomerular filtration rate).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage II (Grade A or B) periodontitis (according to AAP 2017 classification).
* Age range: 20 to 70 years.
* No pathological tooth mobility.
* No furcation involvement caused by periodontal disease.
* No systemic diseases affecting periodontal or renal health.
* No systemic antibiotic use within the previous 3 months.
* No periodontal treatment within the previous 6 months

For Chronic Kidney Disease (CKD) Patients:

* Confirmed CKD diagnosis for at least 3 years (by a consultant nephrologist).
* Receiving conservative management (pre-dialysis).

Exclusion Criteria:

- Stage III or IV periodontitis.

* Grade C periodontal disease.
* Bone loss in more than 10 sites.
* Pathological tooth mobility (Grade II or III).
* Furcation involvement due to periodontal disease.
* Tooth loss due to periodontal disease.
* Heavy smoking (>10 cigarettes/day).
* Pregnancy or lactation.
* Patients undergoing dialysis.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Cystatin C levels after periodontal therapy | Baseline (before treatment) and 4 weeks after completion of periodontal therapy
  Comparison of serum Cystatin C concentration (mg/L) between baseline and 4 weeks post non-surgical periodontal treatment (scaling and root planing) in periodontitis patients with and without chronic kidney disease.

OTHER OUTCOMES:
Improvement in periodontal clinical parameters after Non-Surgical therapy. | Baseline measurement (pre-treatment) and 4 weeks post-treatment completion
  Measurement of changes in clinical periodontal parameters (clinical attachment level CAL) at 4 sites per tooth, 4 weeks after non-surgical periodontal therapy (scaling and root planing) in systemically healthy periodontitis patients.
Change in oral health-related quality of life indicators | Baseline measurement (pre-treatment) and 4 weeks follow-up
  Measurement of changes in OHI-s (Oral Hygiene Index simplified) to assess oral health-related quality of life before and after periodontal therapy across all study groups.
Effect of Periodontal Therapy on Renal Markers | Baseline measurement (pre-treatment) and 4 weeks post-treatment completion
  Evaluation of changes in serum cystatin C levels in chronic kidney disease patients (stages 1-3) 4 weeks after non-surgical periodontal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hashm Daoud, Prof, Study Chair — Tishreen University, faculty of Dentistry; Nebras Naddaf, Phd's student, Principal Investigator — Tishreen University, faculty of Dentistry
Locations (1):
- Tishreen University - faculty of Dentistry, Latakia, Syria